CLINICAL TRIAL: NCT00343629
Title: Bioequivalency Study of Sulindac in Capsule vs. Tablet Formulations
Brief Title: Sulindac Capsules Compared With Sulindac Tablets in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000473167; MAYO-03-1-BIO; MAYO-CPN0576; MAYO-05-004233
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2006-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Sulindac

INTERVENTIONS:
Drug: sulindac
Other: pharmacological study

SUMMARY:
RATIONALE: Giving healthy volunteers sulindac capsules or sulindac tablets may help doctors learn which form of the drug may be more effective in preventing cancer.

PURPOSE: This randomized clinical trial is studying sulindac capsules to see how well they work compared with sulindac tablets in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the systemic exposure of sulindac tablets vs sulindac capsules in healthy volunteers.

Secondary

* Compare the terminal half-life and time of peak drug concentration of sulindac tablets vs sulindac capsules.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive one sulindac capsule followed 7-10 days later by one sulindac tablet.
* Arm II: Participants receive one sulindac tablet followed 7-10 days later by one sulindac capsule.

Blood is collected periodically during treatment for pharmacokinetic studies.

After completion of study therapy, participants are followed at 7-10 days.

PROJECTED ACCRUAL: A total of 28 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy volunteer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hemoglobin ≥ 12.0 g/dL (women)
* Hemoglobin ≥ 13.5 g/dL (men)
* WBC > 3,000/mm³
* Platelet count > 100,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Alkaline phosphatase ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* ALT ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 30 mL/min
* No history of allergic reactions or hypersensitivity to sulindac or other NSAIDs, including aspirin-sensitive asthma or urticaria
* No condition that interferes with ingestion or absorption of oral medications
* No cancer within the past 3 years except nonmelanomatous skin cancer, localized prostate cancer, carcinoma in situ of the cervix, or superficial bladder cancer that was previously treated > 6 months ago
* No uncontrolled concurrent illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction in the past 6 months
  * Chronic renal disease
  * Chronic liver disease
  * Hypertension that is difficult to control
  * Psychiatric illness or social situations that would limit study compliance
* No other significant clinical disorder or laboratory finding that would preclude study participation
* No consumption of alcoholic or caffeinated beverages for ≥ 24 hours prior to study drug administration and until all blood samples have been drawn
* Willing to provide required biologic specimens

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior investigational agents
* More than 6 months since prior regular use of (defined as a frequency of 7 consecutive days for > 3 weeks or > 21 days total) or other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX)-2 inhibitors including, but not limited to, the following:

  * Ibuprofen
  * Ketoprofen
  * Naproxen
* More than 6 weeks since prior oral corticosteroids
* More than 30 days since prior and no concurrent use of any of the following:

  * Methotrexate
  * Corticosteroids
  * Warfarin
  * Ticlopidine
  * Clopidogrel
  * Low molecular weight heparins
  * Abciximab
  * Dipyridamole
  * Eptifibatide
  * Tirofiban
  * Lithium
  * Cyclosporine
  * Hydralazine
  * Angiotensin-converting enzymes (ACE) inhibitors

    * ACE-receptor antagonists allowed
  * Angiotensin-receptor blockers
  * Ginkgo
  * Ketorolac
  * Levofloxacin
  * Loop diuretics
  * Meadowsweet
  * Selective serotonin reuptake inhibitors
  * Danaparoid
* No concurrent regular aspirin use unless prescribed by a physician for prevention

  * A maximum of one aspirin (81 mg/day) allowed
* No concurrent herbal products (e.g., saw palmetto or Hypericum perforatum [St. John's wort])

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2006-04; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Limburg, MD, MPH, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States